CLINICAL TRIAL: NCT03900624
Title: Ideal Steroids for Asthma Treatment in the PICU (iSTAT PICU): A Prospective, Comparative, Single-arm Study Assessing Dexamethasone Versus Methylprednisolone in Severe Status Asthmaticus Admitted to the Pediatric Intensive Care Unit
Brief Title: Ideal Steroids for Asthma Treatment in the PICU
Acronym: iSTAT PICU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00187813
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Results first posted 2022-08-26 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Asthma Childhood
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Single Arm Treatment Group with a Prospective, Comparative Cohort Receiving Standard Care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylprednisolone Arm (No Intervention): Non-randomized, prospective, observational arm of children receiving standard care for status asthmaticus in the PICU with intravenous methylprednisolone.
- Dexamethasone Arm (Experimental): Non-randomized, open-label, prospective use of intravenous dexamethasone for children admitted to the PICU with status asthmaticus.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Non-randomized, open-label, prospective use of intravenous dexamethasone for children admitted to the PICU with status asthmaticus
  Arms: Dexamethasone Arm

SUMMARY:
Determine if differences in (1) pediatric intensive care unit length of stay, (2) continuous nebulized albuterol duration, and (3) a composite outcome of advanced asthma therapy incidence including use of non-invasive ventilation (NIV), terbutaline, inhaled helium and mechanical ventilation between cohorts of children admitted with status asthmaticus to the PICU treated with either IV dexamethasone (DM) or methylprednisolone (MP).

DETAILED DESCRIPTION:
As the pathophysiology of an acute asthma exacerbation is dysregulated inflammatory pathways, standard treatment includes the prompt initiation of intravenous systemic corticosteroids. Corticosteroids reduce the production of many mediators involved in the inflammatory process and inhibit macrophages, monocytes, T-lymphocytes, eosinophils, and basophils, which are activated during this process. Furthermore, corticosteroids improve the efficacy of beta-2 agonists, such as albuterol, a nebulized medication used for bronchodilation in acute asthma exacerbations. There remains an ongoing dialogue among the expert medical community regarding the superiority of specific IV corticosteroid, dosing, route and delivery. This debate continues secondary to a lack of definitive comparative data in the literature. While the benefits of receiving systemic corticosteroids has been demonstrated in multiple studies, to date, no head-to-head trials have been conducted comparing IV systemic corticosteroids in the PICU setting (DM vs. MP).

While several systemic corticosteroids are FDA approved for the treatment of asthma exacerbation including prednisone, prednisolone, MP and DM, the standard practice in PICU-level care is IV MP every 6 hours until enteral medications can be safely tolerated. Recent data from emergency room literature would suggest there is equipoise in use of dexamethasone as an alternative for methylprednisolone due to its increased glucocorticoid (anti-inflammatory) potency. Steroid agents are chosen at the discretion of clinical providers based upon a child's capacity to tolerate enteral medications and the specific clinical setting (outpatient vs. general inpatient vs. critical inpatient).

The investigators have performed a retrospective study over a 2-year period to assess if differences in clinical outcomes or adverse events exist in cohorts defined by DM exposure in the ER. Their data revealed no differences, but most children were switched to MP during their PICU stay making data analyses severely confounded by exposure to the defining characteristics of the comparative cohort. The investigators seek to first prospectively consent individuals to receive DM during their PICU asthma treatment and compare outcomes to PICU asthmatics concurrently admitted to the PICU receiving local standard care (MP). Johns Hopkins All Children's Hospital (JHACH) admits approximately 150 asthmatics per year in the PICU and the investigators hope to enroll up to 50 subjects into a DM only arm. The comparative standard care arm will be assessed at the end of the study period. Primary outcomes include (1) PICU Length of Stay, (2) Continuous nebulized albuterol duration, and (3) a composite outcome including use of non-invasive ventilation (NIV), terbutaline, inhaled helium, inhaled anesthetic gas, mechanical ventilation, and extracorporeal life support. This research will provide the needed epidemiologic and basic comparative data required to power and conduct a definitive, head-to-head trial of DM vs. MP.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are children 5 to 17 years of age with primary admission diagnoses of acute asthma exacerbation or status asthmaticus admitted to the PICU

Exclusion Criteria:

* children with existing tracheostomy, cystic fibrosis, and pulmonary hypertension

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2019-04-21 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony A Sochet, MD, MS, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor IK, Shaw RJ. The mechanism of action of corticosteroids in asthma. Respir Med. 1993 May;87(4):261-77. doi: 10.1016/0954-6111(93)90022-r. No abstract available. PMID 9728226
- [Background] Svedmyr N. Action of corticosteroids on beta-adrenergic receptors. Clinical aspects. Am Rev Respir Dis. 1990 Feb;141(2 Pt 2):S31-8. PMID 1968733
- [Background] Scarfone RJ, Fuchs SM, Nager AL, Shane SA. Controlled trial of oral prednisone in the emergency department treatment of children with acute asthma. Pediatrics. 1993 Oct;92(4):513-8. PMID 8414819
- [Background] Connett GJ, Warde C, Wooler E, Lenney W. Prednisolone and salbutamol in the hospital treatment of acute asthma. Arch Dis Child. 1994 Mar;70(3):170-3. doi: 10.1136/adc.70.3.170. PMID 8135557
- [Background] Storr J, Barrell E, Barry W, Lenney W, Hatcher G. Effect of a single oral dose of prednisolone in acute childhood asthma. Lancet. 1987 Apr 18;1(8538):879-82. doi: 10.1016/s0140-6736(87)92857-1. PMID 2882288
- [Background] Gleeson JG, Loftus BG, Price JF. Placebo controlled trial of systemic corticosteroids in acute childhood asthma. Acta Paediatr Scand. 1990 Nov;79(11):1052-8. doi: 10.1111/j.1651-2227.1990.tb11382.x. PMID 2267922
- [Background] Kattan M, Gurwitz D, Levison H. Corticosteroids in status asthmaticus. J Pediatr. 1980 Mar;96(3 Pt 2):596-9. doi: 10.1016/s0022-3476(80)80872-9. PMID 7359263
- [Background] Keeney GE, Gray MP, Morrison AK, Levas MN, Kessler EA, Hill GD, Gorelick MH, Jackson JL. Dexamethasone for acute asthma exacerbations in children: a meta-analysis. Pediatrics. 2014 Mar;133(3):493-9. doi: 10.1542/peds.2013-2273. Epub 2014 Feb 10. PMID 24515516
- [Background] Paniagua N, Lopez R, Munoz N, Tames M, Mojica E, Arana-Arri E, Mintegi S, Benito J. Randomized Trial of Dexamethasone Versus Prednisone for Children with Acute Asthma Exacerbations. J Pediatr. 2017 Dec;191:190-196.e1. doi: 10.1016/j.jpeds.2017.08.030. PMID 29173304

RESULTS

PARTICIPANT FLOW:
Groups:
- Methylprednisolone Arm - Standard Care: Non-randomized, prospective, observational arm of children receiving standard care for status asthmaticus in the PICU with intravenous methylprednisolone 0.5mg/kg/dose every 6-hours for 5-days.
- Dexamethasone Arm - Interventional Arm: Non-randomized, open-label, prospective use of intravenous dexamethasone 0.25 mg/kg/dose every 6 hours for 2-days for children admitted to the PICU with status asthmaticus.
  Dexamethasone: Non-randomized, open-label, prospective use of intravenous dexamethasone for children admitted to the PICU with status asthmaticus
Period: Overall Study
Arm/Group | Methylprednisolone Arm - Standard Care | Dexamethasone Arm - Interventional Arm
Started | 61 | 31
Completed | 61 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Methylprednisolone Arm - Standard Care: Non-randomized, prospective, observational arm of children receiving standard care for status asthmaticus in the PICU with intravenous methylprednisolone.
- Dexamethasone Arm - Interventional Arm: Non-randomized, open-label, prospective use of intravenous dexamethasone for children admitted to the PICU with status asthmaticus.
  Dexamethasone: Non-randomized, open-label, prospective use of intravenous dexamethasone for children admitted to the PICU with status asthmaticus
- Total: Total of all reporting groups
Arm/Group | Methylprednisolone Arm - Standard Care | Dexamethasone Arm - Interventional Arm | Total
Number analyzed (Participants) | 61 | 31 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.7 (3.8) | 9.3 (3.5) | 9.6 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 13 | 43
  Male | 31 | 18 | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
NHLBI Asthma Classification [Count of Participants; unit: Participants] — National Heart Lung and Blood Institute Chronic Asthma Severity Classification
  Participants
    Intermittent | 10 | 4 | 14
    Mild Persistent | 13 | 7 | 20
    Moderate Persistent | 26 | 10 | 36
    Severe Persistent | 12 | 10 | 22
Pediatric Asthma Severity Score [Median (Inter-Quartile Range); unit: units on a scale] — Score ranges from 5-15. Greater scores signify greater severity of illness with respect to asthma exacerbation.
  units on a scale | 11 [9 to 12] | 10.5 [8 to 12] | 11 [8 to 12]

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay
Description: Hospital length of stay measured in days.
Time Frame: From enrollment through hospital discharge, up to 1 week
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Methylprednisolone Arm - Standard Care | Dexamethasone Arm - Interventional Arm
Number analyzed (Participants) | 61 | 31
days | 2.9 [2.1 to 4] | 2.9 [1.8 to 4.1]
Statistical Analysis 1: Comparison: Methylprednisolone Arm - Standard Care vs Dexamethasone Arm - Interventional Arm; Test type: Superiority; p = 0.632, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Duration of Continuous Nebulized Albuterol
Description: Duration (in days) of continuous nebulized albuterol.
Time Frame: From enrollment through hospital discharge, up to 1 week
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Methylprednisolone Arm - Standard Care | Dexamethasone Arm - Interventional Arm
Number analyzed (Participants) | 61 | 31
days | 1 [0.5 to 1.9] | 0.8 [0.5 to 1.7]
Statistical Analysis 1: Comparison: Methylprednisolone Arm - Standard Care vs Dexamethasone Arm - Interventional Arm; Test type: Superiority; p = 0.725, Wilcoxon (Mann-Whitney)

3. Other Pre Specified Outcome: Number of Participants Receiving an Adjunctive Asthma Therapy
Description: Number of participants receiving an adjunctive therapy:
  * use of non-invasive ventilation (NIV)
  * terbutaline
  * inhaled helium
  * inhaled anesthetic gas
  * mechanical ventilation
  * extracorporeal life support
Time Frame: From enrollment through hospital discharge, up to 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Methylprednisolone Arm - Standard Care | Dexamethasone Arm - Interventional Arm
Number analyzed (Participants) | 61 | 31
Participants | 41 | 16
Statistical Analysis 1: Comparison: Methylprednisolone Arm - Standard Care vs Dexamethasone Arm - Interventional Arm; Test type: Superiority; p = 0.725, Wilcoxon (Mann-Whitney)

4. Other Pre Specified Outcome: Corticosteroid-related Adverse Events
Description: Rates of known corticosteroid-related adverse events including clinically-relevant gastrointestinal bleeding, gastritis, ventilator associated pneumonia, necrotizing enterocolitis, hypertension, hyperglycemia, altered mentation (including hallucinations and delirium), and adrenal insufficiency observed prior to hospital discharge.
Time Frame: From enrollment through hospital discharge, up to 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Methylprednisolone Arm | Dexamethasone Arm
Number analyzed (Participants) | 61 | 31
Participants
  Hyperglycemia | 7 | 2
  Hypertension | 1 | 1
  Adrenal insufficiency | 2 | 0
  Altered mentation | 2 | 0
  Clinically-relevant gastrointestinal bleeding | 0 | 0
  Gastritis | 0 | 0
  Necrotizing enterocolitis | 0 | 0
  Ventilator associated pneumonia | 0 | 0

ADVERSE EVENTS:
Time Frame: From enrollment to hospital discharge or 30-days; whichever comes first.
Arm/Group | Methylprednisolone Arm - Standard Care | Dexamethasone Arm - Interventional Arm
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/31
Other Adverse Events (participants affected / at risk) | 12/61 | 3/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylprednisolone Arm - Standard Care (N=61) | Dexamethasone Arm - Interventional Arm (N=31)
Hyperglycemia (Endocrine disorders) | 7 (7) | 2 (2) — Steroid induced hyperglycemia
Hypertension (General disorders) | 1 (1) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 2 (2) | 0 (0)
Altered Mentation (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT03900624/Prot_SAP_000.pdf